CLINICAL TRIAL: NCT04110418
Title: Methylene Blue Versus Vasopressin Analogue for Treatment of Septic Shock in Preterm Neonate
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rabab Gameel Abd EL hamid allam, Assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWA000017586
Record Dates: First submitted 2019-09-26; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Neonatal Sepsis; Refractory Shock
Keywords: methylene blue; terlipressin; septic shock; preterm neonate
MeSH Terms: conditions — Neonatal Sepsis; Shock; Shock, Septic | interventions — Methylene Blue; Terlipressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylene Blue group (Group MB) (Active Comparator): Methylene Blue is supplied in 1 ml or 10 mL single-dose ampules. Each 1 mL ampule contains 10 mg of methylene blue as a clear dark blue solution
  * Any unused product or waste material should be disposed of in accordance with local practice,
  * For administration to be diluted before use in a solution of 50 mL 5% Dextrose in Water (D5W) in order to avoid local pain, particularly in the paediatric population. Use the diluted solution immediately after preparation.
  * Do not mix with sodium chloride 9 mg/mL (0.9%) solution for injection, because it has been demonstrated that chloride reduces the solubility of methylene blue.
  Interventions: Drug: Methylene Blue
- Terlipressin Group (Group TP ) (Placebo Comparator): The active substance is terlipressin acetate. Each ampoule contains
  1 mg of terlipressin acetate in 8.5 ml solution for injection. This is equivalent to 0.12 mg terlipressin acetate per ml.
  * The powder is to be dissolved in the enclosed solvent and slowly administered intravenously. Further dilution up to 10 ml with sterile isotonic sodium chloride solution is possible.
  * Store in a refrigerator at 2-8˚C.
  * Keep the ampoules in the outer carton in order to protect from light
  Interventions: Drug: Methylene Blue

INTERVENTIONS:
Drug: Methylene Blue — Methylene Blue group (Group MB):will receive IV MB initiated with a first loading dose ( 1 mg/kg over 30 minutes ) then continuous IV infusion( 0.15 mg/kg per hour for up to 24 hours)
  Terlipressin Group (Group TP) Terlipressin will be initiated with a loading dose ( 2 μg/kg intravenous over 30 minutes ) followed by continuous IV infusion starting by 2 μg/kg/h escalating up every 15 minutes up to 20 μg/kg/h
  Other Names: terlipressin acetate

SUMMARY:
A randomized, prospective study comparing methylene blue versus terlipressin in treatment of catecholamines resistant shock in preterm neonate

DETAILED DESCRIPTION:
The study will be an un-blinded, Phase 2, randomized, 1:1, prospective trial comparing methylene blue versus terlipressin in treatment of preterm neonate with catecholamines resistant septic shock the outcome as regard elevation of mean arterial blood pressure will be measured within 72 hours

ELIGIBILITY:
Neonate with Gestational age at birth ≤ 36weeks

Inclusion Criteria:

* diagnosis of Septic shock according to clinical sepsis score of Tollner and Hematologic Scoring System of Rodwell
* Refractory septic shock defined as hypotension although adequate fluid resuscitate and high dose vasopressor(NE >0.5 mcg/kg/min)
* consent form

Exclusion Criteria:

* known case of G6pd deficiency
* Hx of drug allergy MB, NE, terlipressin
* Patients with severely impaired renal function.
* History of maternal drug intake of selective serotonin reuptake inhibitors,and Serotonin-Norepinephrine Reuptake Inhibitors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-02-19 (Estimated); Study Completion 2020-02-19 (Estimated)

PRIMARY OUTCOMES:
to assess the efficancy of each intervention in improving hemodymaic status: time taken to reach adequate mean blood pressure | 24hours
  The time taken to reach adequate mean blood pressure
  Reduction in the dosage of the standard inotropic support

SECONDARY OUTCOMES:
to assess the effect of intervention on survival | 4 days
  mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: rabab allam, physician, Principal Investigator — ain shams university faculty of medicine
Locations (1):
- Neonatal Intensive Care Units (NICUs), Ain Shams University, Cairo, Abbasia, Egypt